CLINICAL TRIAL: NCT03810482
Title: Pedometers and Walking Tests for Pulmonary Hypertension Patients: a First, Prospective Psychology and Concordance Study
Brief Title: Pedometers and Walking Tests for Pulmonary Hypertension Patients
Acronym: HTAPODO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL18_0186
Record Dates: First submitted 2019-01-17; First posted 2019-01-18 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Hypertension, Pulmonary
Keywords: health related quality of life; anxiety; depression; coping; fatigue
MeSH Terms: conditions — Hypertension, Pulmonary; Anxiety Disorders; Depression; Fatigue

STUDY DESIGN:
Intervention Model Description: In this first study, the links between variables and discordance between walking test and pedometer results will be searched.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The study population (Experimental): The study population as described by eligibility criteria.
  Intervention: 6 minute walking test Intervention: pedometer
  Interventions: Device: Pedometer; Other: 6 minute walking test

INTERVENTIONS:
Device: Pedometer — A pedometer will be worn by the patient at home for days 1 to 14 and 60 to 74.
Other: 6 minute walking test — Performed according to current recommendations during routine visits (baseline and ~90 days for the purposes of this study).

SUMMARY:
Concordance between walking tests and pedometer data may seem like a logical outcome for pulmonary hypertension (PH) patients. However, many individuals have discordant results: results much worse or better during an in-hospital walking test as compared to real life activity.

The primary objective of this study is: to determine variables associated with discordance between the distance walked during an in-hospital 6-minute walking test (6MWT) and the average distance travelled per day (observed over a period of 28 days (2 × 14 days) using a pedometer) among PH patients.

DETAILED DESCRIPTION:
Secondarily, the discordance between 6MWT results versus total pedometer recorded distance and versus maximum daily pedometer-recorded distance will be similarly studied. The aim of the study is also to search for variables associated with progression free survival. The relationships between pedometer data and self-reported dyspnea variation will be studied. Factorial analysis may be used to study the overall view of variable correlations and patient similarity/dissimilarity.

ELIGIBILITY:
Inclusion Criteria:

* Patient with idiopathic pulmonary hypertension (PH), familial PH, or PH associated with various pathologies (groups I to IV of the international classification)
* New York Heart Association (NYHA) severity classes II to IV
* Incident cases, or prevalent cases with stable disease over the last 3 months
* Collection of informed written consent
* Affiliation with or beneficiary of a social security program (health insurance)
* Outpatient consulting at the hospital on the day of inclusion
* 6 minute walking test on day of inclusion

Exclusion Criteria:

* Patients protected or unable to give consent according to Article L1121-8 of the French Public Health Code (CSP)
* Pregnant or lactating women according to article L1121-5 of the CSP
* Vulnerable persons according to article L1121-6 of the CSP
* Simultaneous participation in any other research protocol
* It is impossible to correctly inform the patient (language barrier, etc.)
* The patient has already been included in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-03-21 (Actual); Primary Completion 2024-06-21 (Estimated); Study Completion 2024-06-21 (Estimated)

PRIMARY OUTCOMES:
The patient's discordance category as precisely defined here: | 74 days
  Linear regression is performed for the distance walked during an initial 6 minute walking test (6MWT) and the average distance walked per day according to the pedometer intervention. The residuals from this regression will determine categories:
  Category 1 (pedometer high): the 25% of subjects not in category 2 and with higher values for pedometer data
  Category 2 (concordance): the 50% of included subjects with the smallest residuals in terms of absolute value.
  Category 3 (6MWT high): the 25% of subjects not in category 2 and with higher values for 6MWT data

SECONDARY OUTCOMES:
Health related quality of life questionnaire (the Medical Outcome Study - Short Form (SF36)) | Day 0
  This scale evaluates social, emotional and physical health of the patient through 11 questions.
Health related quality of life questionnaire (the Medical Outcome Study - Short Form (SF36)) | Month 3
  This scale evaluates social, emotional and physical health of the patient through 11 questions.
Hospital Anxiety and Depression (HAD) scale | Day 0
  It is a questionnaire which detects if the patient is anxious or depressed through 14 questions.
Hospital Anxiety and Depression (HAD) scale | Month 3
  It is a questionnaire which detects if the patient is anxious or depressed through 14 questions.
State-Trait Anxiety Inventory (STAI) questionnaire | Day 0
  The State-Trait Anxiety Inventory is a 20 question-scale. For each question 4 levels of response are possible from 1 (never) to 4 (always).
State-Trait Anxiety Inventory (STAI) questionnaire | Month 3
  The State-Trait Anxiety Inventory is a 20 question-scale. For each question 4 levels of response are possible from 1 (never) to 4 (always).
Multidimensional Fatigue Inventory (MFI)-20 questionnaire | Day 0
  This questionnaire assesses the severity of the patient fatigue through 20 questions. For each question, 4 levels of response are possible : from "not at all" to "completely".
Multidimensional Fatigue Inventory (MFI)-20 questionnaire | Month 3
  This questionnaire assesses the severity of the patient fatigue through 20 questions. For each question, 4 levels of response are possible : from "not at all" to "completely".
Coping with Health Injuries and Problems Scale | Day 0
  This questionnaire assesses how the patient responds to health injuries and problems with 32 questions. For each question 5 levels of response are possible from 1 (not at all) to 5 (always).
Coping with Health Injuries and Problems Scale | Month 3
  This questionnaire assesses how the patient responds to health injuries and problems with 32 questions. For each question 5 levels of response are possible from 1 (not at all) to 5 (always).

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Bourdin, MD, PhD, Study Director — University Hospitals of Monpellier
Locations (1):
- Arnaud de Villeneuve Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No